CLINICAL TRIAL: NCT06407089
Title: Effectiveness of a Telerehabilitation Program Based on Specific Neck Exercises in Patients With Forward Head Posture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Pilar Pardos Aguilella, Doctor of Physical Therapy, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: C.I. PI24/164
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-05

CONDITIONS: Forward Head Posture; Neck Pain
Keywords: telerrehabilitation; deep cervical muscles; neck muscles; exercise therapy; specific neck exercises
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spinertial Group (SG) (Experimental): Endurance training program of deep cervical flexors and deep cervical extensors with Spinertial device for treatment.
  Endurance training program of deep cervical flexors and deep cervical flexors with Spinertial device for treatment.
  Interventions: Other: Spinertial Group
- Control Group (CG) (No Intervention): The subject continues activities of daily living without intervention.

INTERVENTIONS:
Other: Spinertial Group — Endurance training program of deep cervical flexors and deep cervical extensors with Spinertial device for treatment.
  Endurance training program of deep cervical flexors and deep cervical flexors with Spinertial device for treatment.
  Arms: Spinertial Group (SG)

SUMMARY:
The aim of this study is to compare the effects of a 12-session telerehabilitation program based on Specific Neck Exercises (SNE) with Spinertial to a control group on range of motion, cervical proprioception, and posture in subjects with forward head posture, post-intervention, after one month of follow-up, and after two months of follow-up.

DETAILED DESCRIPTION:
Epidemiological evidence suggests that a sedentary lifestyle is associated with various musculoskeletal conditions, including neck pain. Sedentary behavior during work hours is closely linked to the craniovertebral angle (CVA). Forward head posture, associated with increased vertebral load, predisposes individuals to early onset of degenerative changes, cervical pain, and disability, as well as decreased endurance and strength of the cervical musculature.

Patients with cervical pain may exhibit various clinical manifestations, including weakness of the deep cervical musculature, reduced cervical range of motion (ROM), and cervical disability. Numerous pathologies are described to manifest with localized pain in the cervical region, as well as weakness of the deep cervical musculature and reduced craniovertebral angle (CVA). Examples include cervicogenic dizziness, cervicogenic headache, tension headache, cervical radiculopathy, cervical instability, or chronic mechanical cervicalgia.

The sensorimotor control system is a crucial component of the cervical spine. The deep musculature of the cervical region contains a large number of neuromuscular spindles and mechanoreceptors, providing information about the movement of the head and enhancing dynamic stability during neck movements. The density of neuromuscular spindles in the deep musculature is particularly high, suggesting a significant role in the fine motor control of the cervical spine. Impairment of cervical posture, decreased craniovertebral angle (CVA), proprioception, and alterations in the sensorimotor control system associated with neck pain contribute to recurrence and chronicity.

ELIGIBILITY:
Inclusion Criteria:

* Forward head posture (craniovertebral angle less than 50º).
* Deep flexor strength deficit in craniocervical flexion test.
* Deep extensor strength deficit in neck extensor muscle endurance.
* ≤ 14 score in Neck Disability Index.

Exclusion Criteria:

* Have received cervical treatment during the last six months.
* Presence of any red flag, neurological, or cognitive impairment (inability to - - understand the questionnaires or examination).
* Have received cervical manual therapy treatment during the last six months.
* History of cervical trauma or surgery during the last year.
* Chronic neck pain occurring during the last six months (intensity: visual analogue scale >3/10, frequency >2 days/week, duration >3 hours/day).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Mean Change in Craniovertebral angle (CVA) from baseline | Baseline and 6 weeks, 10 weeks, 14 weeks
  The examiners assess the cranio-vertebral angle (CVA), reflecting the forward head posture position, is the acute anglecreated between the horizontal plane and the line from the tip of the C7 spinous process to the tragion. Head postureis measure as the acute angle between the horizontal plane and the line from the corner of the eye to the tragion(ETH).
Mean Change in Cervical Spine Range of Motion (ROM) from Baseline. | Baseline and 6 weeks, 10 weeks, 14 weeks
  Mean change from baseline in Lower and Upper Cervical Spine Range of Movement (ROM) in the sagittal, frontal and transverse planes after 6 weeks, 10 weeks, and 14 weeks.
  The examiners assess cervical ROM using CROM (Cervical Range-of-Motion Instrument). Cervical flexion, extension, right/left side bending, and right/left rotation will be evaluated in the sagittal, frontal, and transverse planes.
  The examiners assess cervical ROM using CROM (Cervical Range-of-Motion Instrument). Upper cervical flexion, upper cervical extension, and flexion rotation test will be evaluated in the frontal and transverse planes. The flexion rotation test is used to assess the movement of the upper cervical spine and is the most commonly used test in the literature. It is considered positive when there is a decrease of 10 degrees or more in cervical rotation with maximum flexion, in comparison to the contralateral side, or when there is hypomobility of segment C1 with mobility less than 32.
Mean Change in Joint Position error from baseline | Baseline and 6 weeks, 10 weeks, 14 weeks
  Joint Position Error (JPE): The examiners assess the subject's ability (while blindfolded) to relocate the natural head posture (NHP) following the movements of left and right rotation, flexion and extension, upper flexion and upper extension. The relocation error (joint position error, JPE) is the difference between the starting position and the NHP after movement.

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Pardos-Aguilella, Principal Investigator — Universidad de Zaragoza
Locations (1):
- Élite Fisioterapia, María Montessori 2., Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No